CLINICAL TRIAL: NCT01949844
Title: Artifact-Free High-resolution Myocardial Perfusion MRI in Subjects With Abnormal Nuclear Myocardial Perfusion Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel S. Berman (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Daniel S. Berman, Chief, Cardiac Imaging / Nuclear Cardiology, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 28466
Record Dates: First submitted 2013-09-11; First posted 2013-09-25 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease; CAD
Keywords: MRI; Magnetic Resonance Imaging; myocardial perfusion; myocardial perfusion imaging; Novel MRI Techniques
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson; gadoversetamide; Gadolinium; gadolinium compound P760; Magnetic Resonance Imaging; Perfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Suspected coronary artery disease (CAD) (Other): This pilot study has a single arm/group of subjects with suspected CAD based on the following inclusion criteria:
  1. Prior nuclear myocardial perfusion scan (PET/SPECT) with a visual interpretation of definitely abnormal, or prior myocardial infarction; or,
  2. Clinically stable individuals with suspected coronary artery disease on the basis of coronary angiography.
  The study protocol involved only a myocardial perfusion MRI procedure for detection of ischemia (perfusion deficits) using an improved protocol with the administration of a vasodilator drug (Regadenoson/Lexiscan®) and gadolinium-based MRI contrast agent (Optimark®; dose: 0.2 mmol/kg). Lexiscan® was used off-label as a vasodilator drug during the MRI scan (0.4 mg/5mL) supplied by the manufacturer, Astellas Pharma U.S.
  Interventions: Drug: regadenoson; Drug: Optimark®; Device: Myocardial perfusion MRI

INTERVENTIONS:
Drug: regadenoson — Lexiscan® is being used off-label. The FDA Issued IND # is 119898. For the cardiac MRI, Lexiscan® will be used at the same dosage and administration as prescribed in the package insert - 5 mL (0.4 mg regadenoson) as packaged and supplied by the manufacturer, Astellas Pharma U.S., in single-use pre-filled syringes administered by rapid intravenous injection, followed immediately by saline flush.
  Other Names: Lexiscan®
Drug: Optimark® — For the cardiac MR, the contrast agent, Optimark® is administered as a bolus peripheral intravenous injection at a dose of 0.2 mL/kg (0.1 mmol/kg) and at a rate of 1 to 2 mL/sec delivered by manual injection.
  Other Names: gadoversetamide; gadolinium; MRI contrast agent; gadolinium contrast
Device: Myocardial perfusion MRI
  Other Names: magnetic resonance imaging; ischemia; cardiac blood flow; perfusion

SUMMARY:
This is a pilot study in a patient population with suspected coronary artery disease (CAD) as defined by the presence of a prior abnormal nuclear (PET/SPECT) myocardial perfusion scan. In this study design, PET/SPECT will serve as the comparative standard for presence of myocardial ischemia. We intend to determine the accuracy of an improved magnetic resonance imaging (MRI) technique for detection of myocardial ischemia in subjects with suspected CAD.

This is not a study to specifically evaluate the efficacy or safety of the drugs but rather the diagnostic performance of the improved cardiac MRI procedure.

DETAILED DESCRIPTION:
A total of two imaging protocols will be used as "protocol options" in this study (only one of the protocols will be used for each enrolled subject): (1) "Two-day protocol," which involves MRI of subjects who have had a recent abnormal PET/SPECT study and includes an optional second-day visit; (2) "One-day protocol," which involves the subjects undergoing stress myocardial perfusion SPECT and MRI in the same day.

Two blinded readers will interpret MR and SPECT/PET studies by consensus to assess the presence of perfusion deficits at stress and rest.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated nuclear myocardial perfusion (PET/SPECT) study with mild to moderate ischemia or prior myocardial infarction AND a visual scan interpretation of definitely abnormal AND no intervening revascularization since the prior study; or,
* Clinically stable individuals with suspected or known coronary artery disease on the basis of coronary angiography.

Exclusion Criteria:

* < 18 years of age
* Hypotension (systolic blood pressure <100 mm Hg)
* Significant non-coronary cardiac disease (e.g. severe valvular abnormality, significant cardiomyopathy, etc.)
* Persons unable to successfully pass MRI health and safety screening
* Persons whose renal function test does not meet CSMC standard of care MRI contrast protocol requirements (GFR <45 ml/min based on serum creatinine, age, gender, and ethnicity).
* Subjects with contraindications to or intolerance of regadenoson.
* Persons with an allergy to gadolinium-based contrast.
* Persons with a history of kidney or liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05-16 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Berman, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 subjects with suspected coronary artery disease defined based on prior abnormal nuclear myocardial perfusion (PET/SPECT) scan or prior abnormal coronary angiogram were recruited at Cedars-Sinai Medical Center (CSMC) in Los Angeles, CA.
Pre-assignment Details: This pilot study did not involve evaluation of the efficacy of a drug but rather the diagnostic performance of an improved cardiac magnetic resonance imaging (MRI) technique for detection of myocardial ischemia (presence of perfusion deficits) in subjects with suspected coronary artery disease.
Groups:
- Suspected Coronary Artery Disease (CAD): This pilot study involved a single arm/group of subjects with suspected CAD who all underwent cardiac magnetic resonance imaging (MRI) based on the following inclusion criteria:
  1. Prior nuclear myocardial perfusion (PET/SPECT) scan with a visual interpretation of definitely abnormal, or prior myocardial infarction; or,
  2. Clinically stable individuals with suspected coronary artery disease on the basis of coronary angiography.
  Study Protocol: MRI for detection of perfusion deficits using an improved technique with the administration of a vasodilator drug (Regadenoson) and gadolinium-based MRI contrast agent (with standard dose of 0.2 mmol/kg).
  Vasodilator drug (Regadenoson) used in the study: Lexiscan® (FDA-issued IND# 119898) was used off-label as a vasodilator drug during the cardiac MRI scan as prescribed in the package insert (0.4 mg/5mL bolus followed by saline flush) supplied by the manufacturer, Astellas Pharma U.S., in single-use pre-filled syringes.
Period: Overall Study
Arm/Group | Suspected Coronary Artery Disease (CAD)
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Count of Participants
Groups:
- Suspected Coronary Artery Disease (CAD): This pilot study involved a single arm/group of subjects with suspected CAD who were recruited to undergo an improved cardiac magnetic resonance imaging (MRI) protocol with vasodilator stress (Regadenoson) for detection of myocardial perfusion defects. All subjects were recruited based on the following inclusion criteria: (a) prior nuclear myocardial perfusion (PET/SPECT) scan with a visual interpretation of definitely abnormal, or prior myocardial infarction; or, (b) clinically stable individuals with suspected coronary artery disease on the basis of invasive or noninvasive coronary angiography.
Arm/Group | Suspected Coronary Artery Disease (CAD)
Number analyzed (Participants) | 44
Number analyzed (Count of Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Performance (Specificity and Sensitivity) for Detection of Myocardial Perfusion Deficits on Magnetic Resonance (MR) Images
Description: In this study, the approach is to use nuclear myocardial perfusion (prior PET/SPECT scans for the enrolled patients) as the comparative standard for detection of myocardial ischemia (presence of perfusion deficits). Using this approach, the acquired MR images will be analyzed to determine the diagnostic performance (specificity and sensitivity) of the improved MRI technique for detection of myocardial perfusion deficits.
Time Frame: Baseline only
Population: Patients who did not have diagnostically interpretable MRI data were not analyzed.
Measure: Number; unit: percentage of true cases
Arm/Group | Suspected Coronary Artery Disease (CAD)
Number analyzed (Participants) | 38
percentage of true cases
  diagnostic sensitivity | 95
  diagnostic specificity | 94

ADVERSE EVENTS:
Time Frame: Duration of the visit to the medical center for undergoing the cardiac magnetic resonance imaging study (1 day).
Groups:
- Suspected Coronary Artery Disease (CAD): This pilot study involved a single arm/group of subjects with suspected CAD who were recruited to undergo an improved cardiac magnetic resonance imaging (MRI) protocol with vasodilator stress (Regadenoson) for detection of myocardial perfusion defects. All subjects were recruited based on the following inclusion criteria: (a) prior nuclear myocardial perfusion scan with a visual interpretation of definitely abnormal, or prior myocardial infarction; or, (b) clinically stable individuals with suspected coronary artery disease on the basis of invasive or noninvasive coronary angiography.
Arm/Group | Suspected Coronary Artery Disease (CAD)
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

LIMITATIONS AND CAVEATS:
This pilot study did not have a control/placebo arm and did not involve evaluation of the efficacy of a drug but rather the performance of an improved magnetic resonance imaging (MRI) technique with reduced image artifacts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No